CLINICAL TRIAL: NCT05127122
Title: Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles Infusion Treatment for Acute Respiratory Distress Syndrome: A Phase I/II Clinical Trial
Brief Title: Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles Infusion Treatment for ARDS
Acronym: EXIT-ARDS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change in development plan
Sponsor: Direct Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DB-EF-EXITARDS-0003
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: ARDS, Human
Keywords: ExoFlo; EXIT-ARDS; ARDS; Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles; Direct Biologics
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo Saline (Placebo Comparator): Saline
  Interventions: Other: Saline
- 10mL Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles (Experimental): ExoFlo (Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles)
  Interventions: Drug: Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles
- 15mL Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles (Experimental): ExoFlo (Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles)
  Interventions: Drug: Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles

INTERVENTIONS:
Drug: Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles — Injectable
  Other Names: ExoFlo
  Arms: 10mL Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles; 15mL Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles
Other: Saline — Placebo Saline
  Arms: Placebo Saline

SUMMARY:
To evaluate the safety and efficacy of intravenous(IV) administration of bone marrow mesenchymal stem cell derived extracellular vesicles(EV), ExoFlo, as treatment for Acute Respiratory Distress Syndrome.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of intravenous(IV) administration of bone marrow mesenchymal stem cell-derived extracellular vesicles (EV), ExoFlo, as treatment for Acute Respiratory Distress Syndrome. ExoFlo is also referred to as Investigational Product (IP) throughout the protocol. The duration of the study is 60 days, and the endpoints are as follows:

Primary Endpoint:

1. The incidence of serious adverse events.
2. All-Cause Mortality at 28 days.

Secondary Endpoints:

1. Ventilator-free days at 28days.
2. Improvement in partial pressure of arterial oxygen to fraction of inspired oxygen (PaO2/FiO2) ratio from pre-infusion baseline(Day 0)to Day 7.

The study population will consist of 81 inpatient adult patients between 18 and 85 years of age with moderate to severe ARDS as defined by modified Berlin's criteria. Patients will be randomized via Interactive Response Technology to one of the following 3 treatment arms:

1. PLACEBO: Normal saline 100 mL
2. EXPERIMENTAL: IP 10 mL mixed with Normal Saline 90 mL
3. EXPERIMENTAL: IP 15 mL mixed with Normal Saline 85 mL

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (either by the individual or by the individual's healthcare proxy).
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female aged 18-85.
4. Moderate to severe ARDS as defined by modified Berlin definition (See Section 2.2.1), which includes timing within 1 week of known clinical insult or new or worsening respiratory symptoms; bilateral opacities not fully explained by effusions, or lung collapse; respiratory failure not fully explained by cardiac failure or fluid overload; PaO2/FiO2 ≤ 200 mm Hg.
5. Hypoxia requiring noninvasive oxygen support such as Nasal Cannula (NC), Nonrebreather (NRB), Bilevel Positive Airway Pressure (BIPAP), Continuous Positive Airway Pressure (CPAP), high flow nasal cannula oxygen (HFNC O2) or mechanical ventilation (MV) despite initiating standard of care.
6. If the candidate is either a male or female of reproductive potential, he or she must agree to use of double barrier method of highly effective birth control contraception such as condoms with oral contraceptive pill or choose to remain abstinent if already practicing abstinence during the screening period. The required duration of usage of double barrier method OR maintenance of abstinence must include the time from the beginning of the screening period until 90 days following the last dose of the study treatment.

Exclusion Criteria:

1. Vulnerable populations such as pregnant patients, children, individuals with severe physical or mental disabilities who cannot provide meaningful consent.
2. Active malignancy requiring treatment within the last five years.
3. Major physical trauma in the last 2 days, including motor vehicle accidents, assaults, mechanical falls with sequelae of significant bleeding or craniofacial bruising, and surgeries, such that not one or more injury may be undiagnosed at time of screening.
4. Diagnosis or suspected diagnosis of sepsis without basic microbiology cultures (urinalysis, urine culture, two sets of blood cultures, respiratory culture, at least a standard respiratory viral panel PCR) being collected prior to screening. (Note: Standard respiratory viral panel is defined by at least PCR testing for Adenovirus, Influenza A, Influenza B, Parainfluenza 1-3, Rhinovirus/Enterovirus, and RSV.)
5. Duration of mechanical ventilation exceeds 5 days or 120 hours.
6. Severe pre-existing organ dysfunction prior to admission, as evidenced by being currently listed on one or more organ transplant list, or intermittent Hemodialysis (HD) or Peritoneal Dialysis.
7. Presence of severe hematologic disorder or coagulopathy, such as Disseminated Intravascular Coagulopathy, as evidenced by the activation of a Massive Transfusion Protocols (as defined by the rapid administration of packed Red Blood Cells, Fresh Frozen Plasma and Platelets in fixed ratios, including at least 6 packed Red Blood Cells, within a 24 hour period) within 72 hours or frequent thrombosis of catheters (as specified by replacing 2 catheters or more within a 72 hour period of new placement) within 72 hours.
8. Severe anemia or myelodysplastic syndrome requiring more than 10 units of packed Red Blood Cells transfused within the last 12 months.
9. Patient is currently connected to Extracorporal Membrane Oxygenation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of serious adverse events. | 60 days
Number to patients with All-Cause Mortality at 28 days | 28 days

SECONDARY OUTCOMES:
Ventilator-free days at 28days | 28 days
Change in partial pressure of arterial oxygen to fraction of inspired oxygen (PaO2/FiO2) ratio from pre-infusion baseline(Day 0)to Day 7.PaO2 may be calculated from arterial blood gas (ABG)or imputed from the SpO2daily. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Bill Arana, Study Director — Direct Biologics, LLC

IPD SHARING:
Plan to Share IPD: No